CLINICAL TRIAL: NCT03943537
Title: Effects of Intranasal Insulin on Neuroimaging Markers and Cognition in Patients With Psychotic Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Virginie-Anne Chouinard, MD, Research Psychiatrist, Schizophrenia and Bipolar Disorder Research Program, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019P000664
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Psychosis; Schizophrenia; Schizo Affective Disorder; Bipolar I Disorder
Keywords: Psychosis; Insulin; Brain Metabolism; Cognition
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intranasal Insulin (40 IU) (Experimental): 40 IU Novolin-R insulin will be administered one time using the ViaNase intranasal delivery device.
  Interventions: Drug: Intranasal Insulin

INTERVENTIONS:
Drug: Intranasal Insulin — 40 units Novolin R administered intranasally using ViaNase device.
  Other Names: Novolin R

SUMMARY:
This clinical trial is a single center, single dose study of the acute effects of intranasal insulin on energy metabolism and cognitive function in patients with schizophrenia, schizoaffective and bipolar disorders, compared and healthy controls.

DETAILED DESCRIPTION:
Psychotic disorders are common and severe psychiatric disorders. Despite advances in understanding the pathophysiology of these disorders, more effective and tolerable treatments are still needed. Evidence suggests that energy metabolism is altered in psychotic disorders. The investigators recently developed non-invasive MRI-based techniques to quantify redox balance and ATP generation in the brain. Targeting insulin pathways in the brain may allow for modulating abnormalities in energy metabolism. The investigators seek to examine whether intranasal insulin can modulate energy metabolism and improve cognition in patients with psychotic disorders. The study will use magnetic resonance spectroscopy (MRS) technology to measure in vivo energy metabolism processes in the brain, before and after the administration of intranasal insulin. Investigators will also measure changes in cognition with the administration of intranasal insulin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders (DSM) diagnoses of schizophrenia, schizoaffective disorder or bipolar disorder with psychotic features OR
* Healthy Controls (no history of DSM psychiatric diagnoses, nor history of the same in first-degree relatives)

Exclusion Criteria:

* Psychiatric hospitalization within the last 4 weeks
* Unstable/active disease or potential contraindications, such as liver disease, kidney disease, uncontrolled hypertension, significant or unstable medical illness
* Currently prescribed: antidiabetic agents, including oral antidiabetic medications and insulin, intranasal medication, steroids, weight loss agents
* Pregnant or breast-feeding, not using an effective form of contraception for at least 3 months, and/or not abstinent for 1 month prior to enrollment
* History of significant head injury
* Contraindication to MRI scans (claustrophobia, cardiac pacemakers, metal clips and stents on blood vessels, artificial heart valves, artificial arms, hands, legs, etc., brain stimulator devices, implanted drug pumps, ear implants, eye implants or known metal fragments in eyes, exposure to shrapnel or metal filings, other metallic surgical hardware in vital areas, certain tattoos with metallic ink, certain transdermal patches, metal-containing IUDs).
* Medical conditions preventing blood draws
* History of electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) within the last 3 months
* BMI > 35 or body weight > 350 lbs or BMI <18
* DSM diagnosis of substance use disorder in the past month
* For Healthy Controls:
* Taking medication other than birth control

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginie-Anne Chouinard, M.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with schizophrenia, schizoaffective disorder, or bipolar disorder with psychotic features were recruited from a variety of McLean Hospital outpatient settings, the Registry of Research Participants for the Psychotic Disorders Division, and online advertising methods. A phone screening was conducted before enrollment to assess basic eligibility criteria. Healthy controls were recruited through online advertisements.
Pre-assignment Details: After phone screening, participants were asked to complete an in-person screening visit to confirm study eligibility. The visit included a structured clinical interview (SCID-5) to confirm psychiatric diagnosis, psychiatric scales, blood draw, and medical history interview. Based on the results of these assessments, participants were excluded if they had unstable or active medical problems, diabetes, active substance use disorder, pregnancy, or MRI contraindications.
Groups:
- Patients: Patients with diagnostic and Statistical Manual of Mental Disorders (DSM) diagnoses of schizophrenia, schizoaffective disorder or bipolar disorder with psychotic features. All participants received 40 IU Novolin-R insulin administered one time using the ViaNase intranasal delivery device.
- Controls: Healthy Controls (no history of DSM psychiatric diagnoses, nor history of the same in first-degree relatives). All participants received 40 IU Novolin-R insulin administered one time using the ViaNase intranasal delivery device.
Period: Overall Study
Arm/Group | Patients | Controls
Started | 41 | 46
Completed | 21 | 18
Not Completed | 20 | 28

BASELINE CHARACTERISTICS:
Groups:
- Patients: 21 patients with diagnostic and Statistical Manual of Mental Disorders (DSM) diagnoses of schizophrenia, schizoaffective disorder or bipolar disorder with psychotic features. All participants received 40 IU Novolin-R insulin administered one time using the ViaNase intranasal delivery device.
- Controls: 18 healthy Controls (no history of DSM psychiatric diagnoses, nor history of the same in first-degree relatives). All participants received 40 IU Novolin-R insulin administered one time using the ViaNase intranasal delivery device.
- Total: Total of all reporting groups
Arm/Group | Patients | Controls | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.47 (5.29) | 25.40 (3.64) | 25.44 (4.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 11 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 18 | 12 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 14 | 27
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Brain Redox State
Description: Changes in brain NAD+/NADH ratio as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Patients | Controls
Number analyzed (Participants) | 18 | 16
ratio | -0.269 [-0.769 to 0.231] | -0.485 [-1.077 to 0.107]

2. Primary Outcome: Changes in Brain ATP
Description: Changes in ATP concentration as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: mM
Arm/Group | Patients | Controls
Number analyzed (Participants) | 20 | 17
mM | 0.017 [-0.121 to 0.154] | 0.119 [-0.006 to 0.244]

3. Primary Outcome: Changes in Brain PCr
Description: Changes in Phosphocreatine (PCr) concentration as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: mM
Arm/Group | Patients | Controls
Number analyzed (Participants) | 20 | 17
mM | 0.013 [-0.030 to 0.056] | -0.033 [-0.070 to 0.005]

4. Primary Outcome: Changes in Brain CK
Description: Changes in creatine kinase (CK) enzyme rate as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: s^-1
Arm/Group | Patients | Controls
Number analyzed (Participants) | 20 | 16
s^-1 | 0.009 [-0.012 to 0.029] | 0.006 [-0.012 to 0.025]

5. Primary Outcome: Changes in STROOP Color-word Interference Score
Description: Changes in STROOP assessment color-word condition interference score. This score is calculated as follows, with C being the number of items answered correctly in the color condition, W being the number answered correctly in the word condition, and CW being the number of items answered correctly in the color-word condition: CW - (C x W)/(C+W). Higher scores indicate better cognitive function.
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Patients | Controls
Number analyzed (Participants) | 21 | 18
score on a scale | 1.11 [-0.38 to 2.61] | 0.94 [-0.14 to 2.01]

6. Primary Outcome: Changes in BACS Digit Sequencing Score
Description: Changes in BACS digit sequencing scores, ranging from 0 - 36. Higher scores indicate better cognitive function.
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Patients | Controls
Number analyzed (Participants) | 21 | 18
score on a scale | 0.05 [-0.35 to 0.45] | 0.16 [-0.20 to 0.51]

7. Primary Outcome: Changes in BACS Symbol Coding
Description: Changes in BACS Symbol Coding test, with scores ranging from 0 - 110. Higher scores indicate better cognitive function.
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Patients | Controls
Number analyzed (Participants) | 21 | 18
units on a scale | 0.74 [0.37 to 1.11] | 0.83 [0.58 to 1.09]

8. Primary Outcome: Changes in BACS Verbal Fluency Scores
Description: Changes in BACS verbal fluency subscale z-scores, measured by number of words generated over 60-second trials. A z-score of 0 indicates the population mean. Higher scores indicate better cognitive function.
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: z-score
Arm/Group | Patients | Controls
Number analyzed (Participants) | 21 | 18
z-score | 0.22 [-0.07 to 0.50] | 0.43 [0.14 to 0.72]

9. Secondary Outcome: Changes in Brain pH.
Description: Changes in pH as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: pH
Arm/Group | Patients | Controls
Number analyzed (Participants) | 20 | 17
pH | 0 [-0.007 to 0.007] | -0.004 [-0.012 to 0.003]

10. Secondary Outcome: Changes in Brain Inorganic Phosphate Concentration.
Description: Changes in inorganic phosphate (Pi) concentration as measured by in vivo 31P magnetic resonance spectroscopy
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: mM
Arm/Group | Patients | Controls
Number analyzed (Participants) | 20 | 17
mM | -0.002 [-0.022 to 0.017] | -0.020 [-0.044 to 0.005]

11. Secondary Outcome: Change in Fasting Blood Glucose Levels.
Description: Safety outcome.
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Patients | Controls
Number analyzed (Participants) | 21 | 18
mg/dL | 4.62 [1.35 to 7.89] | 2.17 [0.56 to 3.77]

12. Secondary Outcome: Change in Fasting Blood Insulin Levels.
Description: Safety outcome.
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: uIU/mL
Arm/Group | Patients | Controls
Number analyzed (Participants) | 21 | 18
uIU/mL | 0.110 [-0.634 to 0.854] | -0.228 [-0.877 to 0.421]

13. Secondary Outcome: Change in Brain Glutamate Concentration
Description: Changes in glutamate (Glu) concentration as measured by in vivo proton magnetic resonance spectroscopy
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: mM
Arm/Group | Patients | Controls
Number analyzed (Participants) | 21 | 18
mM | -0.382 [-0.959 to 0.195] | 0.475 [-0.171 to 1.121]

14. Secondary Outcome: Changes in Brain Glutamine Concentration
Description: Changes in glutamine (Gln) concentration as measured by in vivo proton magnetic resonance spectroscopy
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: mM
Arm/Group | Patients | Controls
Number analyzed (Participants) | 21 | 18
mM | -0.110 [-0.296 to 0.075] | 0.105 [-0.132 to 0.342]

15. Secondary Outcome: Changes in Brain Glutathione Concentration
Description: Changes in glutathione (GSH) concentration as measured by in vivo proton magnetic resonance spectroscopy
Time Frame: 6 hours, pre- and post- 40 IU intranasal insulin
Measure: Mean (95% Confidence Interval); unit: mM
Arm/Group | Patients | Controls
Number analyzed (Participants) | 21 | 18
mM | -0.029 [-0.091 to 0.032] | 0.148 [0.032 to 0.263]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected on the day of the intervention visit with one-time intranasal insulin administration.
Arm/Group | Patients | Controls
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/18
Other Adverse Events (participants affected / at risk) | 0/21 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients (N=21) | Controls (N=18)
Nasal irritation (Skin and subcutaneous tissue disorders) | 0 | 1
Headache with nausea after insulin administration (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT03943537/Prot_SAP_000.pdf